CLINICAL TRIAL: NCT00596193
Title: NPY Regulation of Nociceptors in Clinical Inflammation
Brief Title: Neuropeptide Y (NPY) Regulation of Nociceptors
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20010247H
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Pain
Keywords: Hyperalgesia; nociceptors; Neurons
MeSH Terms: conditions — Pain; Hyperalgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: patients with normal or irreversible pulpitis teeth with capsaicin administered at increasing volumes.
- Group II: Patients with normal teeth only with capsaicin added at a specific volume only

SUMMARY:
Neuropeptide Y (NPY) potently inhibits pain neurons in rats, but does this occur in human pain neurons? This hypothesis will be tested using microdialysis probes in patients who elect to have root canal treatment or extraction of thier tooth.

DETAILED DESCRIPTION:
The ongoing studies in rats indicate that a sympathetically-derived neuropeptide, neuropeptide Y (NPY), potently inhibits the activity of the capsaicin-sensative class of nociceptors (i.e., "pain" neurons). It is not know whether these results, generated from rodent studies, occur in human tissues under normal or inflamed conditions. We plan to test the hypothesis that NPY inhibits the initiation of neurogenic inflammation, as measured by reduced release of substance P, from capsaicin-sensitive class of petidergic neurons innervating normal and inflamed dental pulp. Such actions would be physiologically and clinically significant, since inhibition of exocytosis from peripheral terminals of nociceptive primary afferent fibers would likely alter neurogenic inflammation, local vasodilation and , possibly pain. Our research strategy takes advantage of a uniquely innervated tissue: dental pulp. Application of any physiologic stimulus to human dental pulp, including thermal, osmotic, chemical or mechanical, produces only pain. Thus, virtually all sensory neurons that innervate pulp appear to be nociceptors. Accordingly, application of drugs to pulpal sensory neurons targets a population of sensory neurons consisting predominantly of nociceptors.

The research questions are as follows:

1. Determine the capsaicin concentration-response curve from evoking the release of immunioreactive substance P (iSP) from normal and inflamed dental pulp.
2. Determine the effect of NPY on altering basal and capsaisin-evoked release of iSP from normal and inflamed dental pulp.

We will evaluate the hypothesis that NPY inhibits capsaicin-sensitive neurons in humans using microdialysis probes implanted into anesthetized dental pulp, with release of immunoreactive substance P (iSP) as our dependent measure. This study will include patients who have elected to have a root canal procedure performed or to have a tooth extracted.

ELIGIBILITY:
Inclusion Criteria:

* teeth with diagnosis of normal pulp or irreversible pulpitis
* mandibular teeth
* indication for either root canal or extraction of tooth
* age between 18-50

Exclusion Criteria:

* history of taking steroids within the last month
* history of hyperthyroidism, hypertension, asthma, uncontrolled or complicated Type-2 diabetes, drug abuse
* age less than 18 or greater than 50
* maxillary teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental Patients
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2001-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hargreaves, DDS,PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States